CLINICAL TRIAL: NCT00375635
Title: Removal of Protein Bound Uremic Toxins in Chronic Hemodialysis Patients by Modified Plasma Separation and Adsorption Combined With Hemodialysis
Brief Title: Removal of Protein Bound Uremic Toxins by Modified Plasma Separation and Adsorption Combined With Hemodialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: MBD2006
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Last update posted 2006-09-13 (Estimated); Status verified 2006-09

CONDITIONS: Uremia
Keywords: mFPSA; Uremic toxins; Protein bound toxins; Uremia; Chronic hemodialysis
MeSH Terms: conditions — Uremia

INTERVENTIONS:
Procedure: mFPSA treatment

SUMMARY:
The aim of this study is to examine removal of protein bound uremic substances by mFPSA in chronic hemodialysis patients. mFPSA is an extracorporal blood purification system developed for detoxification in acute liver failure by removal of protein bound as well as water soluble substances.

DETAILED DESCRIPTION:
Measurements of uremic protein bound substances before and after mFPSA and a preceding routine hemodialysis session.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Anuria
* Chronic hemodialysis dependence

Exclusion Criteria:

* No present history of bleeding episodes
* Cardiac diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2006-03; Study Completion 2006-10

PRIMARY OUTCOMES:
Blood pressure
Safety serological parameters
Concentrations of protein bound uremic toxins

SECONDARY OUTCOMES:
Bleeding episodes

CONTACTS AND LOCATIONS:
Overall Officials: Mette B Damholt, MD,Ph.d., Principal Investigator — Rigshospitalet P2132; Soren D Ladefoged, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Copenhagen, Denmark